CLINICAL TRIAL: NCT05408728
Title: Dietary Sugar Hyper-absorptive Intestinal Phenotype as a Predictor of Weight Loss Post-bariatric Surgery
Brief Title: Dietary Sugar Absorptive Phenotype for Prediction of Weight Loss Outcome
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dilhana S. Badurdeen, Principal Investigator, Mayo Clinic
Other Study IDs: 22-001407
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obese; Healthy; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obese patients scheduled for Bariatric surgery: Subjects scheduled for Bariatric Surgery (BS) and will receive pre-BS Esophagogastroduodenoscopy (EGD) as a part of your standard care will have biopsies from the small intestine taken during the EGD procedure for this study.
  Interventions: Procedure: Endoscopic biopsy
- Lean controls naive to Bariatric surgery: Subjects presenting for surveillance/screening EGD procedure as part of their standard medical care will have biopsies from the small intestine taken during the EGD procedure for this study.
  Interventions: Procedure: Endoscopic biopsy

INTERVENTIONS:
Procedure: Endoscopic biopsy — Upper small intestinal biopsies from patients undergoing BS will be collected during routine standard of care screening EGD and again from the same patients at 1 year during routine standard of care surveillance EGD (esophageal reflux screening/surveillance). Biopsy-derived enteroid cultures and tissue samples from pre- and one-year post BS will be examined for expression level of sugar transporters and gluconeogenic enzymes; glucose and fructose absorption

SUMMARY:
This study is trying to determine whether the success of bariatric surgery can be predicted by evaluating the dietary sugar absorptive characteristics in the small intestine and if there is any gene expression change on the dietary sugar absorptive characteristics.

ELIGIBILITY:
Inclusion Criteria:

- Obese patients (BMI ≥ 30) scheduled for BS undergoing standard of care screening EGD, or lean BS-naïve individuals (BMI ≤ 25) subjected to EGD for routine clinical indications as part of standard care.

Exclusion Criteria:

* Adults unable to consent, including non-English speakers.
* Pregnant women because endoscopy is a risk factor. All patients of childbearing age undergo history as well as urine pregnancy test as a standard of care prior to undergoing endoscopy as the procedure is performed under anesthesia.
* Prisoners.
* Subjects with preexisting conditions (e.g., bleeding at the time of the procedure, suspected perforation during the standard-of-care procedure) will be excluded from the study at the time of the endoscopy.
* Have a contraindication to endoscopy.
* A history of surgery on the stomach or small intestine.
* Type 1 diabetes (clinical diagnosis and/or positive glutamic acid decarboxylase antibodies).
* Using weight loss medications.
* Active malignancy within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients scheduled for bariatric surgery (BS) (both men and women of any racial/ethnic background), or lean BS-naïve subjects presenting for surveillance/screening endoscopy procedure as part of their standard medical care (controls).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of obese patients with altered dietary sugar hyper-absorptive phenotype after bariatric surgery | 18 months

SECONDARY OUTCOMES:
Epigenetic changes measured in the intestinal mucosa of obese patients with dietary sugar hyper-absorptive phenotype after bariatric surgery | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dilhana Badurdeen, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No